CLINICAL TRIAL: NCT05911971
Title: Specific Upper Airway Reeducation in Moderate Obstructive Sleep Apnea Syndrome: a Randomized Controlled Trial
Brief Title: Upper Airway Reeducation in Moderate Obstructive Sleep Apnea Syndrome
Acronym: SAOSGENIO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP210997; 2021-A02688-33 (Other: IDRCB)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Moderate Obstructive Sleep Apnea Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific reeducation (Experimental): Specific reeducation
  Interventions: Other: Experimental
- Sham comparator (Sham Comparator): Sham reeducation
  Interventions: Other: Sham comparator

INTERVENTIONS:
Other: Experimental — specific reeducation (not detailed to maintain blinding of participants)
  Arms: Specific reeducation
Other: Sham comparator — sham reeducation (not detailed to maintain blinding of participants)
  Arms: Sham comparator

SUMMARY:
The aim of this study is to evaluate the effectiveness of a specific reeducation performed by speech therapists in moderate obstructive sleep apnea syndrome, as an alternative to the continuous Positive Anyway Pressure (CPAP) and the mandibular advancement device.

DETAILED DESCRIPTION:
Patients will be recruited in the sleep pathology department, following a sleep consultation and/or a polysomnography. They will be randomized between 2 reeducation groups (specific reeducation or sham reeducation) and will have to perform their respective exercises during 3 months. Only one of the 2 reeducations is expected to be effective. To limit performance and measure bias, patients will not be aware of the content of the reeducation in the other group (participants partially blinded of study hypothesis) and therefore these are not described in detail here. The initial clinical assessment will be repeated at 3 and 6 months, by assessors blinded to the reeducation arm, in order to evaluate the short and medium term effectiveness on the the Apnea-Hypopnea Index (AHI) and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years old minimum
* Diagnosis of moderate OSAS: AHI ≥ 15 events/h and < 30 events/h at PSG M0
* BMI < 35 kg/m2

Exclusion Criteria:

* MoCA < 26 (Montreal Cognitive Assessment)
* Craniofacial malformations
* Regular use of hypnotic medications
* Untreated hypothyroidism
* Stroke history
* Cardiac insufficiency
* Severe uncontrolled coronary heart disease
* Severe obstructive nasal disease
* Patients with indication for CPAP in first intention
* Pregnant or breastfeeding woman
* Current participation in another interventional research in OSA
* No affiliation to a social security system or legal beneficiary (except AME,Aide médicale d'état)
* Absence of free, informed, written consent
* Contraindications for TMS: intracranial metallic implant, pacemaker and/or recent or severe cardiac disease, epilepsy, vascular, traumatic, tumor, infectious or metabolic brain lesions, severe alcoholism
* Protected adult under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in apnea-hypopnea index (AHI) | between 0 and 3 months after randomization
  Apnea-hypopnea index (AHI) is the number of apnoeas or hypopnoeas per hour of sleep, measured by polysomnography during a minimum 6-hour night of inpatient sleep. Polysomnograms will be interpreted by a blinded somnologist.

SECONDARY OUTCOMES:
Change of the Apnea-Hypopnea Index (AHI) | between 0 and 6 months after randomization
  Apnea-hypopnea index (AHI) is the number of apnoeas or hypopnoeas per hour of sleep, measured by polysomnography during a minimum 6-hour night of inpatient sleep. Polysomnograms will be interpreted by a blinded somnologist.
Change of the MBLF(Bucco-Linguo-Facial Motor Function) score | between 0 and 3 months and between 0 and 6 months after randomization
  Quantitative evaluation of the patient's lingual mobility by the speech therapist. The test consists of the execution of 13 lingual praxias rated from 0 (no contraction) to 3 (normal contraction), with a total score from 0 to 39
Change of the lingual strength | between 0 and 3 months and between 0 and 6 months after randomization
  measured by collecting the maximum pressure in kPa with an tongueometer.
Change of lingual endurance | between 0 and 3 months and between 0 and 6 months after randomization
  Following the same principle as lingual strength, lingual endurance (inversely proportional to fatigability) is measured with a tongueometer by quantifying the duration during which the patient can maintain 50% of his maximum pressure. The target value is then set to 50% of the patient's maximum pressure and the duration (in seconds)
Change of the size of the genioglossus representation in cm² within the motor cortex | between 0 and 3 months after randomization
  by collecting motor evoked potentials of the genioglossus in response to transcranial magnetic stimulation (TMS) applied to the anterolateral region of the right vertex between 0 and 3 months.
Change of quality of life on the SF-36 | between 0 and 3 months and between 0 and 6 months after randomization
  Quality of life will be studied by the SF-36 generalist questionnaire completed by the patient. 36 items divided into 9 dimensions: physical activity, limitations due to physical condition, physical pain, perceived health, vitality, life and relationships with others, psychological health, limitations due to psychological condition, evolution of perceived health. Score from 0 (minimum subjective health) to 100 (maximum subjective health).
Change of sleep quality on the Pittsburgh Sleep Quality Index | between 0 and 3 months and between 0 and 6 months after randomization
  Sleep quality will be studied by the Pittsburgh Sleep Quality Index completed by the patient.19 questions are divided into 7 composite scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, medication use, daytime dysfunctions) ranging from 0 (no difficulty) to 3 (severe difficulty). The global score is calculated by adding the 7 composite scores, the score obtained ranging from 0 to 21. The quality of sleep is investigated over the previous month.
Change of daytime drowsiness on the Epworth Drowsiness Scale | between 0 and 3 months and between 0 and 6 months after randomization
  Daytime drowsiness will be studied by the Epworth Drowsiness Scale completed by the patient. 8 items rated from 0 (no chance of drowsiness) to 3 (systematic drowsiness), total score from 0 to 24. A score greater than or equal to 11 corresponds to daytime sleepiness.
Presence of subjective symptoms , each taken independently | At 3 months and 6 months after randomization
  subjective evaluation by the patient following questions:snoring every night or so (yes/no), high intensity of snoring (heard through a door or complaint from the entourage (yes/no),nocturia (yes/no) if yes frequency of episodes, morning headaches (yes/no),dry mouth at night or upon waking (yes/no),impression of non-restorative sleep (yes/no),bad sleep (yes/no), if yes, number of awakenings per nigh, fatigue (yes/no), daytime sleepiness (yes/no),impatience in the legs (yes/no),nightmares (yes/no), other symptoms (yes/no)
Change of the cervical circumference measurement (at the level of the cricoid) | between 0 and 3 months and between 0 and 6 months after randomization
  in cm, using a tape measure
Change of the respiratory sensation sitting at rest | between 0 and 3 months and between 0 and 6 months after randomization
  Using a visual analogue scale, consisting of a 10 cm plastic ruler graduated in mm presented horizontally. The side presented to the patient has a straight non graduated line, the left end of which corresponds to "no respiratory discomfort" and the right end to "intolerable respiratory discomfort".On the other side, there are millimetre graduations only visible to speech therapist. The position of the cursor chosen by the patient allows to read the intensity of the respiratory discomfort, which is measured in mm
Change of change in respiratory sensation between sitting and full decubitus | between 0 and 3 months and between 0 and 6 months after randomization
  after the measurement of the respiratory sensation while sitting at rest, the patient is put in complete decubitus and the change of his respiratory discomfort between these 2 positions is measured. This change is collected using a visual analog scale, consisting of a 10 cm plastic ruler graduated in mm presented horizontally. The side presented to the patient has a straight, non-scaled line with "maximum aggravation" at the left end to "maximum improvement" at the right end, with a central marker to indicate "no change". On the other side, there are millimeter graduations only visible to speech therapist. The position of the cursor chosen by the patient allows to read the intensity of the respiratory discomfort, the results are expressed as a percentage of the full scale, the latter being defined as the distance between the central marker and one of the extremities, with a "+" sign for improvement and a "-" sign for worsening which is measured in mm.
Change of sleep latency | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of N3 latency | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the paradoxical sleep latency | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
change of sleep efficiency | between 0 and 3 months and between 0 and 6 months after randomization
  calculated as total sleep time (TST) versus time from sleep to wakefulness (TWA), during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the total sleep time (TST) | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the length of the N1 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the percentage (related to the TST) of the N1 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in percentage of TST, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the length of the N2 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the percentage (related to the TST) of the N2 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in percentage of TST, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the length of the N3 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the percentage (related to the TST) of the N3 | between 0 and 3 months and between 0 and 6 months after randomization
  measured in percentage of TST, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the length of paradoxical sleep | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the percentage (related to the TST) of paradoxical sleep | between 0 and 3 months and between 0 and 6 months after randomization
  measured in percentage of TST, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the length of intrasleep vigil | between 0 and 3 months and between 0 and 6 months after randomization
  measured in minutes, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the percentage (related to the TST) of intrasleep vigil | between 0 and 3 months and between 0 and 6 months after randomization
  measured in percentage of TST, during polysomnography in a minimum 6-hour night of inpatient sleep
Change of the index of micro-awakenings | between 0 and 3 months and between 0 and 6 months after randomization
  Is the number of micro-awakenings per hour of sleep, measured by polysomnography during a minimum 6-hour night of inpatient sleep.
Change of the index of micro-awakenings of respiratory origin | between 0 and 3 months and between 0 and 6 months after randomization
  Is the number of micro-awakenings of respiratory origin per hour of sleep, measured by polysomnography during a minimum 6-hour night of inpatient sleep.
Change of the number of periodic leg movements | between 0 and 3 months and between 0 and 6 months after randomization
  Is the number of periodic leg movements per hour of sleep, measured by polysomnography during a minimum 6-hour night of inpatient sleep.
Change of number of sleep cycles | between 0 and 3 months and between 0 and 6 months after randomization
  Is the number of sleep cycle, measured by polysomnography during a minimum 6-hour night of inpatient sleep.
Compliance with treatment | at 3 months
  declared by the patient via the logbook given to the patient at the initial assessment. After each exercises session, the patient will have to complete the day, indicate the time spent and any difficulties encountered. Telephone follow-up of compliance will be carried out by the speech therapist or the clinical study technician every month. Compliance will be evaluated by the percentage of days when the patient will have declared to have carried out exercises for a duration higher than 50% of the theoretical duration of the exercises session

CONTACTS AND LOCATIONS:
Overall Officials: Diane PICARD-DUBOIS, Principal Investigator — APHP
Locations (1):
- Service des pathologies du sommeil, Pitié-Salpêtrière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.